CLINICAL TRIAL: NCT03346629
Title: Evaluating the Safety, Acceptability and Feasibility of an Outpatient "Day Procedure" Service Documenting the Roles of Health Workers in the Provision of Medical Abortion at 13-18 Weeks Gestation
Brief Title: Outpatient Service for Mid-trimester Termination of Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: CREHPA (Unknown); Kathmandu Medical College and Teaching Hospital (Other); Kathmandu Model Hospital (Unknown); KIST Medical College (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1039
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Abortion in Second Trimester
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mifepristone + Misoprostol (Experimental): Intervention: 200mg mifepristone followed 24-48 h later with 400mcg misoprostol (repeat Q3)
  Interventions: Drug: Mifepristone + Misoprostol

INTERVENTIONS:
Drug: Mifepristone + Misoprostol — A single dose of 200 mg mifepristone (one tablet) to be taken orally either at home or at the hospital, followed 24-48 hours later with 400mcg misoprostol (buccal) at home. The participant will return to the hospital one to two hours after taking the initial dose of misoprostol to receive repeated doses of 400 mcg misoprostol until the abortion occurs.

SUMMARY:
This study seeks to evaluate the safety, acceptability and feasibility of an outpatient "day procedure" for medical abortion at 13-18 weeks gestation. The study regimen will consist of a single dose of 200 mg mifepristone to be taken orally either at home or at the hospital, followed approximately 24 - 48 hours later with administration of 400 mcg misoprostol. Repeat doses of 400 mcg (two tablets) of misoprostol will be administered buccally every three hours until the abortion is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Have an ongoing pregnancy of 13-18 weeks gestation
* Meet legal criteria to obtain an abortion at 13-18 weeks gestation (legal criteria include pregnancy resulting from rape or incest, fetal malformation and/or if the pregnancy affects the physical or mental health of the woman)
* Has access to a phone where she can be reached at the 2-week follow-up
* Be willing to follow study procedures

Exclusion Criteria:

* Known allergy to mifepristone or misoprostol/prostaglandin or other contraindications to the use of mifepristone or misoprostol
* Any contraindications to vaginal delivery
* More than one prior cesarean delivery
* Living more than 2 hours away from the hospital

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Successful medical abortion | 0 - 48 hours after first dose of mifepristone
  Proportion of women who have a successful medical abortion without recourse to surgical intervention and return home on the same day as misoprostol induction

SECONDARY OUTCOMES:
Induction-to-abortion interval | 0 - 48 hours after first misoprostol dose
  Median time elapsed between administration of the first misoprostol dose until expulsion of both fetus and placenta
Total dose of misoprostol | 0 - 48 hours after first misoprostol dose
  Average number of doses of misoprostol
Safety - Proportion of participants who experience at least one of the following: extramural delivery, hemorrhage requiring transfusion, infection, uterine rupture, prolonged hospitalization, any complications | 2 weeks after initial visit
  Proportion of participants who experience at least one of the following: extramural delivery, hemorrhage requiring transfusion, infection, uterine rupture, prolonged hospitalization, any complications
Tasks performed by certified staff | 0 - 72 hours after receipt of mifepristone
  Type of task performed (i.e. counseling, monitoring vital signs, administering drugs, monitoring woman's condition, post-abortion contraception, managing discharge)
Hospital admission time | Within 0 - 48 hours after the second dose of misoprostol
  Average total hospital admission time
Side Effects | 0 - 48 hours after first dose of misoprostol
  Proportion of participants experiencing side effects (severity incidence, and severity of pain based on a 0-10 point scale)
Initiation-to-abortion interval | 0 - 72 hours after receipt of mifepristone
  Median time elapsed between administration of the mifepristone dose until expulsion of both fetus and placenta

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Blum, MPH, Principal Investigator — Gynuity Health Projects; Monica Dragoman, MD, MPH, Principal Investigator — Gynuity Health Projects; Chanda Karki, MD, Principal Investigator — Kathmandu Medical College; Dina Abbas, MPH, Principal Investigator — Gynuity Health Projects; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Anand Tamang, MPhil, Principal Investigator — CREHPA
Locations (3):
- Nepal (3):
  - KIST Medical College, Teaching Hospital, Imadol, Lalitpur
  - Kathmandu Medical College, Kathmandu
  - Kathmandu Model Hospital, Kathmandu